CLINICAL TRIAL: NCT01759030
Title: Double Blind Randomized Clinical Study Evaluating Efficacy and Safety of BCD-020 and MabThera in Patients With Rheumatoid Arthritis Who Had an Inadequate Response or Intolerance to Other DMARDs Including One or More TNF Inhibitor Therapies
Brief Title: Study of Safety and Efficacy of BCD-020 Comparing to MabThera in Patients With Rheumatoid Arthritis
Acronym: BIORA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIORA (BCD-020-2)
Record Dates: First submitted 2012-12-20; First posted 2013-01-02 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis, DMARDs; rituximab; biosimilar; interchangeability
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MabThera (F. Hoffmann-La Roche Ltd.) (Active Comparator): Stage 1 (week 1 - week 24) MabThera will be administered at a dose of 1000 mg, IV (on day 1 and day 15).
  Stage 2 (week 24 - 48) If the disease activity remains on Week 24 the patient will undergo the second randomization (1:1 ratio): if he/she randomised into group A then he/she recieves BCD-020 at a dose f 1000 mg, IV, once in 2 weeks, 2 infusions per course (on day 1 and day 15); if he/she if he/she randomised into group B then he/she continues to recieve MabThera at a dose f 1000 mg, IV, once in 2 weeks, 2 infusions per course (on day 1 and day 15).
  MabThera/BCD-020 will be used in combination with methotrexate (irrespectively to study stage).
  Interventions: Drug: Rituximab
- BCD-020 (CJSC BIOCAD) (Experimental): Stage 1 (week 1-week 24) BCD-020 will be administered at a dose of 1000 mg, IV (on day 1 and day 15).
  Stage 2 (week 24-48) If the disease activity remains on Week 24 the patient will undergo the second randomization (1:1 ratio): if he/she randomised into group A then he/she recieves MabThera at a dose f 1000 mg, IV, on day 1 and day 15; if he/she if he/she randomised into group B then he/she continues to recieve BCD-020 at a dose f 1000 mg, IV, on day 1 and day 15.
  MabThera/BCD-020 will be used in combination with methotrexate (irrespectively to study stage).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Patients will will receive rituximab a dose of 1000 mg , intravenously, slowly, once in 2 weeks, with 2 infusions per course (on day 1 and day 15).
  Other Names: MabThera, Rituxan, BCD-020

SUMMARY:
The purpose of this study is to prove that efficacy, safety and immunogenicity of BCD-020 is equivalent to MabThera when used in combination with methotrexate for the treatment of patient with rheumatoid arthritis

DETAILED DESCRIPTION:
This is an international multicenter double-blind randomized clinical study of the efficacy and safety (Phase III) with an active comparator; the study provides the additional evaluation of the interchangeability of rituximab biosimilar and original product MabThera.

The study will include 308 subjects with active seropositive rheumatoid arthritis who had intolerance or inadequate response to current therapy regimens including one or more TNF inhibitors, or who had contraindications to TNF inhibitors.

The first 24-week stage includes one course of rituximab therapy. The first study stage proposes central randomization into 2 large groups (1:1): patients from the first group will recieve BCD-020 (rituximab manufactured by CJSC BIOCAD) at a dose 1000 mg in a drop-wise manner on day 1 and day 15; patients from the second group will recieve MabThera at a same regimen.

On the final visit of Stage 1 (visit 11 at week 24) all efficacy parameters must be evaluated. If the disease activity remains (DAS28 score ≥2.6 or increased by 0.6 points or more compared to the last measurement) the patient will recieve another course of rituximab treatment. In this case a partial crossover (Stage 2) will take place (by means of the second randomization): one half of patients with active RA, previously treated with BCD-020, will receive MabThera at a dose 1000 mg on day 1 and day 15; and one half of patients with active RA, previously treated with MabThera, will receive BCD-020 at a dose 1000 mg ion day 1 and day 15. After the first rituximab infusion performed for retreatment, the patient will undergo 24-week follow-up (counted starting from the date of retreatment initiation). Thus, effects of the switch from BCD-020 to MabThera and vice versa will be assessed in 24 weeks after the crossover (Stage 2 of the study).

Patients in whom remission of RA (DAS28 < 2.6) is reported on week 24 counting from the initial randomization will undergo the follow up for the next 24 weeks. During this period they will attend 3 visits (weeks 32, 40 and 48) in order to monitor the disease. If the exacerbation occurs within the time period not corresponding to week 32 or week 40, the patient will be invited to the study site for an out-of-schedule visit. If disease exacerbation is confirmed, he/she undergoes the second randomization, second rituximab treatment course and further follow up for 6 months (as described above).

ELIGIBILITY:
Inclusion Criteria:

* Having signed a written informed consent form.
* Patients must be from 18 to 80 years of age (both ages inclusive)
* Rheumatoid arthritis confirmed according to ACR 1987 criteria.
* Seropositive rheumatoid arthritis.
* Active rheumatoid arthritis during the last 3 months.
* Disease score according to DAS28 of 3.2 or more, TJC≥8 (68), SJC≥8 (66), hsCRP≥6 mg/l, ESR≥28 mm/hr (by Westergren) at the moment of screening.
* Patient's functional status - class I-III according to ACR classification
* Inadequate response to DMARDs that include one or more TNF inhibitors, intolerance or contraindications to TNF inhibitors.
* Necessity of methotrexate treatment during the last 4 weeks prior to screening period with stable/consistent dosage of 7.5 - 20 mg per week.
* Patient's ability (in Investigator's opinion) to follow the protocol procedures;
* Willingness to use contraception during all study period.

Exclusion Criteria:

* Patients with Felty's syndrome (irrespectively to clinical form).
* Patient's functional status - class IV according to ACR classification .
* Rheumatoid arthritis low activity (less than 3.2 according to DAS28).
* Concomitant therapy:

  * Previous treatment with any biological drug products causing CD20+ lymphocyte depletion, including biological investigational drugs.
  * Treatment with azathioprine within 28 days before the study initiation and with leflunomide within 8 weeks before the study's principal phase (treatment with rituximab).
  * Intra-articular glucocorticosteroids within 4 weeks before the study's principal phase (treatment with rituximab).
  * Necessity for prednisone or its equivalent administration at dose more than 10 mg per day.
  * Necessity for prednisone or its equivalent administration at dose ≤10 mg per day in cases when this dose wasn't stable/consistent during last 4 weeks.
  * Necessity for administration of non-steroidal anti-inflammatory drugs for arthritis treatment in cases when its doses were not stable/consistent during last 4 weeks.
* Pregnancy and breast-feeding.
* Changes of laboratory values:

  * Hemoglobin level is less than 100 g/l;
  * Leucocyte level is less than 3,0×10e9/l;
  * Absolute neutrophil count is less than 1,5×10e9/l;
  * Thrombocyte level is less than 100×10e9/l.
* Confirmed chicken pox within 30 days before inclusion to the screening.
* Confirmed herpes zoster infection.
* Acute forms of any infectious diseases, history of chronic infections with severe clinical manifestations.
* Active tuberculosis, history of latent tuberculosis.
* Inflammatory disease of the joints (present or in anamnesis) not related to rheumatoid arthritis (including gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease and others) or other systemic autoimmune disease (including systemic lupus erythematosus, Crohn's disease, ulcerative colitis, systemic scleroderma, inflammatory myopathy, mixed forms of connective tissue inflammatory diseases, cross-syndrome and others).
* Juvenile idiopathic arthritis or juvenile rheumatoid arthritis and/or rheumatoid arthritis developed before the age of 16.
* Any determined immunodeficiency.
* Pernicious anemia.
* Confirmed cobalamine deficiency.
* Other somatic diseases (apart from rheumatoid arthritis) that can increase the probability of adverse events during the study or can influence the estimation of symptom manifestation of RA ; mask, enhance or alter the symptoms of RA or cause clinical or laboratory symptoms similar to that of RA;
* Positive results of serological test of Hepatitis B surface antigen (HbsAg) or presence of Hbc IgM together with positive results of HBV PCR test, presence of antibodies to Hepatitis C virus, syphilis or HIV.
* Major surgery within 28 days prior to the trial principal phase (treatment with rituximab).
* Any mental disorder, including major depression and/or suicidal thoughts in anamnesis that can, in Investigator's opinion, create a risk for the patient or influence the patient's ability to follow the study protocol.
* Unstable angina pectoris.
* Myocardial infarction within less than 1 year prior to participation in the study.
* Severe central or peripheral nervous system diseases.
* Drug addiction, alcoholism.
* Known hypersensitivity to murine proteins or any other components of the medications used in the treatment, methotrexate, folic acid and any drugs used in premedication.
* Presence of malignant neoplasm, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ and any malignancy with complete remission of more than 5 years;
* Simultaneous participation in any other clinical trial, as well as former participation in other clinical trials within 3 months before this study initiation; previous participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2012-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who have reached ACR20 within 24 weeks after the treatment initiation | week 24

SECONDARY OUTCOMES:
Frequency of adverse events (AE) and serious adverse events (SAE) that is related, in Investigator's opinion, to rheumatoid arthritis therapy | during all time of participation in the study
Frequency of AE and SAE grade 3-4 that is related, in Investigator's opinion, to rheumatoid arthritis therapy | during all time of participation in the study
Number of cases of early withdrawal from the study caused by AE or SAE | during all time of participation in the study
Level of binding and neutralizing antibodies to rituximab in patients from both groups | at screening, week 12, week 24
CD19+ and CD20+ lymphocyte counts | before infusion, after the 1st and the 2nd infusion of rituximab, on day 3,17,29 after the 1st infusion, at week 12,24,48

OTHER OUTCOMES:
CD3+ lymphocyte count | before infusion, after the 1st and the 2nd infusion of rituximab, on day 3,17,29, at week 12,24,48
Number of patients in each group who have reached ACR20 | week 48
Number of patients in each group that have reached ACR50/70 | week 24, week 48
Number of patients in each group with low RA activity according to DAS28 | week 24, week 48
Number of patients in each group with RA remission according to DAS28 | week 24, week 48
Number of patients in each group with RA remission according to ACR/EULAR | week 24, week 48
X-ray characteristic of the involved joints | week 24, week 48
  1. Rate of progression in structural joint damage in Total Modified Sharp Score (erosion score, joint space narrowing score);
  2. Percentage of patients without radiologic progression (by Steinbrocker).
Functional ability index according to HAQ | week 12, week 24, week 48
Quality of life assessment by SF-36 questionnaire | week 12, week 24, week 48
Level of hsCRP and ESR by Westergren | Day 29, weeks 8,12,16,20,24,32,40,48
Serum levels of IgA, IgG, IgM | Day 17,29, 46 weeks 24,48
Serum level of rituximab | 0 h, 3 h, 6 h after infusion, on day 3 (48 h after the 1st infusion), day 17 (48 hours after the 2nd infusion), day 29 (after 336 hours after the 2nd infusion) and day 46 (744 hours after the 2nd infusion)
Hazard ratio for the absence of remission according to DAS28 after 24 weeks from the switching from MabThera to BCD-020, comparing to the patients, which were retreated with MabThera without the switching to BCD-020 | 48 weeks
Hazard ratio for the absence of remission according to DAS28 after 24 weeks from the switching from BCD-020 to MabThera, comparing to the patients, which were retreated with BCD-020 without the switching to MabThera | 48
Percentage of patients in each group that have reached ACR20/50/70 within 24 weeks after the retreatment initiation | 48 weeks
Percentage of patients in each group with low RA activity according to DAS28 (2.6-3.2) in 24 weeks after the retreatment initiation | 48 weeks
Percentage of patients in each group with RA remission according to DAS28 (<2.6) in 24 weeks after the retreatment initiation | 48 weeks
Percentage of patients in each group with RA remission according to ACR/EULAR 2011 in 24 weeks after the retreatment initiation | 48 weeks
Radiography characteristic of the involved joints after 24 weeks from the retreatment initiation including | 48 weeks
Functional disability index according to HAQ-DI after 24 weeks from the start of retreatment | 48 weeks
Quality of life assessment by SF-36 questionnaire after 24 weeks from the start of retreatment | 48 weeks
Percentage of patients in each group withf binding and neutralizing antibodies to rituximab at screening, at week 12 an week 24 after the first infusion during the first cycle of therapy and after 24 weeks from the start of retreatment | 48 weeks
Mean titre of binding and neutralizing antibodies to rituximab at screening, at week 12 and week 24 after the first infusion during the first cycle of therapy and after 24 weeks from the start of retreatment | 48 weeks
Hazard ratio of any AE, that is related, in Investigator's opinion, to the use of rituximab and which has occurred after the switching from MabThera to BCD-020, in comparison with patients who were retreated with MabThera without switching to BCD-020 | 48 weeks

CONTACTS AND LOCATIONS:
Locations (40):
- Belarus (4):
  - Gomel Regional Clinical Hospital, Homyel
  - City Clinical Hospital №1, Minsk
  - City Clinical Hospital №9, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- India (23):
  - Satellite Orthopaedic Hospital & Research Centre Pvt Ltd, Ahmadābād
  - Smt NHL Medical College and SethVS General Hospital, Ahmadābād
  - Government Medical College and Hospital Panchakki Road, Aurangabad
  - Bangalore Medical College and Research Institute, Victoria Hospital, Bangalore
  - Pristine Hospital and Research Center Pvt. Ltd, Bangalore
  - Sapthagiri Institute of Medical Sciences and Research Centre#15, Bangalore
  - Sri Venkateshwara Hospital, Bangalore
  - Sri Ramachandra Medical Centre, No.1, Chennai
  - Swami Vivekananda National Institrute of Rehabilitation Training and research, Cuttack
  - Gandhi Hospital, Department of Orthopedics, Hyderabad
  - Sri Sri Holistic Hospitals, Hyderabad
  - Sumana Hospitals, Research Department, Hyderabad
  - Yashoda Hospital, Hyderabad
  - Jaipur Hospital, Lal Kothi, Near SMS Stadium, Jaipur
  - SMS Medical College & Hospital, Jaipur
  - Calcutta national medical college, Kolkata, Kolkata
  - Bhatia Hospital, Medical Research Society, Mumbai
  - Government Medical College and Hospital, Nagpur
  - Jawarlal Institute of Postgraduation Medical Education and Research, Puducherry
  - B.J Medical college Sassoon General Hospital, Near Pune Railway Station, Pune
  - Medipoint Hospitals Pvt Ltd, Pune
  - Ruby Hall Clinic, Pune
  - Christian Medical College, Vellore
- Russia (10):
  - Chelyabinsk Regional Clinical hospital, Chelyabinsk
  - Clinical Hospital at Chelyabinsk Railway Station, Chelyabinsk
  - Kursk regional hospital, Kursk
  - Research Institute of Rheumotology, Moscow
  - Nizhegorodskaya Regional Clinical Hospital named after N.A. Semashko, N.Novgorod
  - Limited liability company Consultation and Diagnostic Center "Zdorovyye sustavy", Novosibirsk
  - North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg
  - Local hospital at the station Smolensk OAO RZD, Smolensk
  - Smolensk State Medical Academy, Smolensk
  - Novgorod regional clinical hospital, Veliky Novgorod
- Ukraine (3):
  - Kharkiv City Clinical Emergency Hospital n.a. O.I.Meschaninov, Kharkiv
  - National Research Center "Cardiology Institute n.a. M.D.Strazheska", Kyiv
  - Odessa Regional Cardiology Dispensary, Odesa